CLINICAL TRIAL: NCT07353203
Title: Safety and Efficacy of Hip Assist Powered Exoskeleton for Gait Training in Patients With Late Subacute and Chronic Stroke, Multi-center, Randomized Controlled Pilot Study
Brief Title: Safety and Efficacy of Hip Assist Powered Exoskeleton for Gait Training in Patients With Late Subacute and Chronic Stroke
Acronym: brain disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-08-147
Record Dates: First submitted 2025-12-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Stroke; Subacute Stroke; Exoskeleton

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gait assistance mode group (Experimental): Gait training is performed in gait assistance mode while wearing a hip-assist powered exoskeleton
  Interventions: Device: gait assistance mode group
- Resistance mode (Experimental): Gait training is performed in Resistance mode while wearing a hip-assist powered exoskeleton
  Interventions: Device: Resistance mode

INTERVENTIONS:
Device: gait assistance mode group — A total of 10 sessions of gait training were performed using the hip-assist powered exoskeleton for 5 weeks (30 minutes per session)
  Arms: gait assistance mode group
Device: Resistance mode — A total of 10 sessions of gait training were performed using the hip-assist powered exoskeleton for 5 weeks (30 minutes per session)
  Arms: Resistance mode

SUMMARY:
The aim of this study is to evaluate the safety of gait training using a hip-assist powered exoskeleton. This will be assessed by collecting all device-related adverse events occurring during the entire intervention period, which consists of a total of 10 sessions within 5 weeks across two different gait rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 85 years.
2. Patients with hemiplegia resulting from ischemic or hemorrhagic stroke.
3. Patients in the late subacute or chronic phase, with stroke onset of 3 months or more (in cases of recurrent stroke, based on the most recent event). Functional Ambulation Category (FAC) score of 3 or higher.
4. Patients capable of safely wearing the hip-assist powered exoskeleton and using it with minimal assistance.

   * Height: 140 cm - 190 cm
   * Weight: 80 kg or less
5. Patients who were capable of independent walking and had no disability in daily self-care activities prior to stroke onset (based on the last stroke for recurrent patients). (mRS ≤2)
6. Patients who have received approval for study participation from the attending medical staff.

Exclusion Criteria:

1. Severe cognitive impairment (Mini-Mental State Examination [MMSE] < 10) or severe speech impairment/aphasia.
2. History of major orthopedic surgery, such as hip, knee, or ankle arthroplasty, within the last 3 months.
3. Fractures, open wounds, or unhealed ulcers in the lower extremities.
4. Patients for whom gait training with the powered orthopedic device is difficult due to severe medical conditions, such as cardiovascular or pulmonary diseases.
5. History of osteoporotic fractures.
6. Patients with other neurological diseases affecting gait (e.g., Parkinson's disease, multiple sclerosis, etc.).
7. Any other cases where the investigator deems participation in the study to be inappropriate.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
10 Meter Walk Test | Baseline, after 5 intervention sessions(week 3) , and after 10 intervention sessions(Week 5)
  (lower limb motor score in 10 Meter Walk test at post-intervention) - (lower limb motor score in 10 Meter Walk Test at baseline) Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea